CLINICAL TRIAL: NCT03497598
Title: Preventing Recurrent Urinary Tract Infections With α-D-mannose: a Prospective, Randomized, Double-blinded Placebo-controlled Trial
Brief Title: Preventing Recurrent Urinary Tract Infections With α-D-mannose
Acronym: PUTIM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: not enough patients
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Gloria Ryu, Assistant medical director, Kantonsspital Aarau
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PUTIM
Record Dates: First submitted 2018-04-05; First posted 2018-04-13 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Urinary Tract Infections
Keywords: D-mannose
MeSH Terms: conditions — Urinary Tract Infections | interventions — Mannose; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mannose (Experimental): 2g d-mannose (white) powder (Hänseler AG, Herisau, Switzerland) daily (sachet) for 6 months.The powder is dispensed in neutral sticks and ready to be dissolved in 100ml of water for oral Ingestion.
  rUTI diary
  Interventions: Drug: Mannose
- placebo (Placebo Comparator): 2g Hänseler lactose (white) powder (Hänseler AG, Herisau, Switzerland) daily (sachet) for 6 months. The powder is dispensed in neutral sticks and ready to be dissolved in 100ml of water for oral Ingestion.
  rUTI diary
  Interventions: Drug: Lactose

INTERVENTIONS:
Drug: Mannose — The powder is dispensed in 2g neutral sticks and ready to be dissolved in 100ml of water for daily oral ingestion.
  Other Names: D-Mannose Oral Powder
  Arms: mannose
Drug: Lactose — The powder is dispensed in 2g neutral sticks and ready to be dissolved in 100ml of water for daily oral ingestion.
  Other Names: Lactose powder
  Arms: placebo

SUMMARY:
In this trial, women with history of recurrent urinary tract infections (UTIs) will be followed over the course of 6 months. The women will be randomized either to D- Mannose or Placebo.

The primary objective of this study is to investigate if treatment with D-mannose reduces the risk for a UTI recurrence compared to treatment with Placebo.

H0: Women with history of recurrent UTIs treated with D-Mannose on average have the same number of recurrent UTIs over the course of 6 months compared to women treated with Placebo.

H1: Women with history of recurrent UTIs treated with D-Mannose on average have fewer recurrent UTIs over the course of 6 months compared to women treated with Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Women
* ≥ 3 UTIs within the last 12 months or ≥ 2 UTIs within the last 6 months;
* Laboratory urine culture: <103 CFUs
* Age > 18 years

Exclusion Criteria:

* UTIs ≥ 12 within 1 year
* Pregnancy or Lactation
* Immune disease
* Lactose intolerance
* Urinary tract anomaly
* Systemic infection
* Newly started hormone therapy within the last 6 months
* Antibiotic prophylaxis within the last 6 months
* α-D-mannose intake within the last month
* Use of catheters
* Diabetes mellitus
* Participation to other studies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Frequency of UTIs | 6 months
  Frequency of UTIs (defined as ≥103 CFU/ 1mL of clean midstream urine) within the 6 months treatment period with D-mannose.

SECONDARY OUTCOMES:
During UTI: Dysuria | during every UTI in the 6 months period
  4 categories: no, mild, moderate, severe
During UTI: Urgency | during every UTI in the 6 months period
  4 categories: no, mild, moderate, severe
During UTI: Frequency | during every UTI in the 6 months period
  4 categories: no, mild, moderate, severe
During UTI: Flank (side) pain | during every UTI in the 6 months period
  4 categories: no, mild, moderate, severe
During UTI: Cystalgia | during every UTI in the 6 months period
  4 categories: no, mild, moderate, severe
During UTI: Back pain | during every UTI in the 6 months period
  4 categories: no, mild, moderate, severe

OTHER OUTCOMES:
Presence/absence of E. coli, Enterococcus faecali, Klebsiella pneumoniae, Streptococcus agalactiae, Proteus mirabilis, Citro-bacter freundii, Pseudomonas aeruginosa, others not specified | at the screening and during every UTI in the 6 months period
  2 categories: yes, no
Weight | at the screening
  in kilograms
Height | at the screening
  in cm
Menopause status | at the screening
  3 categories: premenopausal, perimenopausal, postmenopausal
Sexual activity | at the screening
  2 categories: yes, no
Medication | at the screening and during every UTI in the 6 months period
  2 categories: yes, no if yes: Name of the medication, dosage, reason for medication, start and end date of medication
Age | at the screening
  in years
Birth control | at the screening
  2 categories: yes, no
Number of CFU | at the screening and during every UTI in the 6 months period
  number

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Ryu, MD, Principal Investigator — Kantonsspital Aarau
Locations (1):
- Kantonsspital Aarau, Aarau, Switzerland

REFERENCES:
- [Background] Kranjcec B, Papes D, Altarac S. D-mannose powder for prophylaxis of recurrent urinary tract infections in women: a randomized clinical trial. World J Urol. 2014 Feb;32(1):79-84. doi: 10.1007/s00345-013-1091-6. Epub 2013 Apr 30. PMID 23633128
- [Background] Domenici L, Monti M, Bracchi C, Giorgini M, Colagiovanni V, Muzii L, Benedetti Panici P. D-mannose: a promising support for acute urinary tract infections in women. A pilot study. Eur Rev Med Pharmacol Sci. 2016 Jul;20(13):2920-5. PMID 27424995
- [Background] Phe V, Pakzad M, Haslam C, Gonzales G, Curtis C, Porter B, Chataway J, Panicker JN. Open label feasibility study evaluating D-mannose combined with home-based monitoring of suspected urinary tract infections in patients with multiple sclerosis. Neurourol Urodyn. 2017 Sep;36(7):1770-1775. doi: 10.1002/nau.23173. Epub 2016 Nov 4. PMID 27813195
- [Derived] Cooper TE, Teng C, Howell M, Teixeira-Pinto A, Jaure A, Wong G. D-mannose for preventing and treating urinary tract infections. Cochrane Database Syst Rev. 2022 Aug 30;8(8):CD013608. doi: 10.1002/14651858.CD013608.pub2. PMID 36041061